CLINICAL TRIAL: NCT01211353
Title: Personalized Drinking Feedback Interventions for OEF/OIF Veterans
Brief Title: Personalized Drinking Feedback Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Matthew P. Martens, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21AA020180-01 (NIH); 1R21AA020180-01 (NIH)
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Alcohol Abuse
Keywords: Alcohol; Brief Intervention; Personalized Feedback; Veterans
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized Drinking Feedback (Experimental): Personalized feedback on drinking behaviors
  Interventions: Behavioral: Personalized Drinking Feedback
- Education-Only (Active Comparator): Educational information about alcohol
  Interventions: Behavioral: Education-Only

INTERVENTIONS:
Behavioral: Personalized Drinking Feedback — Personalized feedback about one's drinking habits
  Arms: Personalized Drinking Feedback
Behavioral: Education-Only — Educational information about alcohol use
  Arms: Education-Only

SUMMARY:
The objective of this research is to better understand how to reduce hazardous drinking among OEF/OIF veterans by assessing the effectiveness of a low-cost, computer-delivered preventative program.

DETAILED DESCRIPTION:
Excessive drinking among OEF/OIF veterans represents an important public health problem for both the veterans themselves and those with whom they interact. The objective of this research is to better understand how to reduce hazardous drinking among this group by assessing the effectiveness of a low-cost, computer-delivered preventative program. It is hypothesized that an intervention that provides personalized feedback about drinking behaviors will be more effective than an education-only control condition at reducing alcohol use and negative alcohol-related consequences.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF Veteran

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Daily Drinking Questionnaire | Past 30 Days
  Several quantity/frequency measures of alcohol use

SECONDARY OUTCOMES:
Short Inventory of Problems | Past 6 Months
  Measures alcohol-related problems

CONTACTS AND LOCATIONS:
Overall Officials: Mattjew P Martens, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Harry S Truman Memorial VA Medical Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No